CLINICAL TRIAL: NCT04534101
Title: Medical Mindfulness: Virtual Reality Mindfulness Therapy for Anxiety and Pain Management in Patients With Acute and Chronic Pain
Acronym: VR Mindfulness
Status: Suspended | Type: Observational
Why Stopped: Temporarily paused due to COVID-19 and expected to resume. Resumption timeline unclear due ongoing pandemic. This is not a suspension of IRB approval.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Linda Nguyen, Clinical Associate Professor, Stanford University
Other Study IDs: 45300
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Acute Pain; Chronic Pain
MeSH Terms: conditions — Acute Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inpatient Subjects: Inpatients will be presented with an informed consent. If they sign the consent, they will then be given a VR headset pre- programmed with content that they may use for the duration of their stay. GI patients headsets will be collected when they are discharged. There are pain and anxiety analog scales at the end of each program. This data will be downloaded to Stanford. Patient's will not be entering their PHI. we will know who has headsets, as they will be numbered. Patient who are hospitalized for chronic pain will be allowed to take the VR headset home for month and be asked to return it at their followup outpatient visit.
  Interventions: Behavioral: Virtual Reality Mindfulness
- Outpatient Subjects: Outpatient: Patient's who are about to undergo gastrointestinal disease testing or be seen for an outpatient GI appointment will be presented with an informed consent. If they sign the consent, they will be given the VR headset to use prior to their procedure. There are pain and anxiety analog scales at the end of each program. This data will be downloaded to Stanford Medicine Box.Patient's will not be entering their PHI. we will know who has headsets, as they will be numbered.
  Interventions: Behavioral: Virtual Reality Mindfulness

INTERVENTIONS:
Behavioral: Virtual Reality Mindfulness — This study is designed to test the feasibility, acceptability and effectiveness of VR mindfulness in patients as they undergo various medical therapies to treat their acute or chronic conditions.

SUMMARY:
Adults and children undergoing medical care (inpatient or outpatient) often experience pain and anxiety either as a result of their medical condition or a side effect of medical procedures. The purpose of this study is to create a registry of patients using virtual reality (VR) mindfulness therapy through different aspects of their medical care to determine if VR mindfulness therapy is more effective than the standard of care (i.e., no technology based distraction) for treating or preventing anxiety and pain in adults and children suffering from chronic pain, GI conditions where pain is a common symptom, or undergoing any painful medical procedure (i.e. IV access, blood draws, endoscopy, surgery). The anticipated primary outcome will be reduction of pain and anxiety for both acute and chronic pain.

DETAILED DESCRIPTION:
Inpatient: Inpatients will be presented with an informed consent. If they sign the consent, they will then be given a VR headset pre- programmed with content that they may use for the duration of their stay. GI patients headsets will be collected when they are discharged. There are pain and anxiety analog scales at the end of each program. This data will be downloaded to Stanford. Patient's will not be entering their PHI. we will know who has headsets, as they will be numbered. Patient who are hospitalized for chronic pain will be allowed to take the VR headset home for month and be asked to return it at their followup outpatient visit.

Outpatient: Patient's who are about to undergo gastrointestinal disease testing or be seen for an outpatient GI appointment will be presented with an informed consent. If they sign the consent, they will be given the VR headset to use prior to their procedure. There are pain and anxiety analog scales at the end of each program. This data will be downloaded to Stanford Medicine Box.Patient's will not be entering their PHI. we will know who has headsets, as they will be numbered.

ELIGIBILITY:
Identify inclusion criteria.

Participants must:

1. be between ages of 5-80 years of age
2. have comprehension of instructions in the English language
3. English speaking
4. Must be able to comprehend ICF
5. Have a medical appointment or procedure at Stanford/LPCH (inpatient or outpatient) that may cause pain or anxiety.

Identify exclusion criteria.

General Exclusion Criteria are as follows:

1. Significant cognitive impairment/developmental delays
2. Seizure Disorder
3. history of motion sickness with virtual reality
4. severe visual impairment

Ages: 5 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Males and females age 5-80 of all ethnic backgrounds. We will enroll from GI outpatient clinics (pediatric and adult) as well as any patients who are hospitilized for acute or chronic pain as well as those who are in the preoperative room getting an IV.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-07-10 (Actual); Primary Completion 2023-07-10 (Estimated); Study Completion 2023-07-10 (Estimated)

PRIMARY OUTCOMES:
VR Mindfulness Acceptability | Up to 1 day (before and after VR use)
  Assess the acceptability of a virtual reality mindfulness meditation tool by patients who are experiencing pain, patients diagnosed with gastrointestinal disorders where pain is a common symptom, and by patients undergoing medical procedures.
Anxiety Outcome | Up to 1 day (before and after VR use)
  Collect patient report outcome data on anxiety before and after using virtual reality mindfulness meditation.
Pain Outcome | Up to 1 day (before and after VR use)
  Collect patient report outcome data on pain levels before and after using virtual reality mindfulness meditation.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Nguyen, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided